CLINICAL TRIAL: NCT03777891
Title: Effect of Silicone Gel Versus Contractubex Phonophoresis for Post-burn Hypertrophic Scars: A Single Blind Randomized Controlled Trial
Brief Title: Effect of Silicone Gel Versus Contractubex Phonophoresis for Post-burn Hypertrophic Scars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, Deputy Director of Quality Assurance Unit, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001870
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Phonophoresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Experimental): received Silicone gel phonophoresis: Silicone gel (strataderm) was applied to the scar then the ultrasound was implemented by the therapist. The ultrasound parameters were set as following, frequency: 1 MHz, intensity: 0.5 W/cm2 and the treatment time was 5 minutes. The Ultrasound Device is Sonopulse 590: Nonius, sonopuls 590, S.NO.03-202 type 14663.900 was a therapeutic ultrasound device manufactured by Enraf Holland.
  Interventions: Combination Product: phonophoresis with different material
- group B (Experimental): received Contractubex phonophoresis: Contractubex (Merz Pharma, Frankfurt, Germany was applied to the scar then the ultrasound was implemented by the therapist. The ultrasound parameters were set as following, frequency: 1 MHz, intensity: 0.5 W/cm2 and the treatment time was 5 minutes.
  Interventions: Combination Product: phonophoresis with different material
- group C (Experimental): received Corticosteroid phonophoresis: A thin film of coupling medium (gel) was put on the hypertrophic scar and sufficient quantity of Triamcinolone was put by a syringe over the whole scar then the ultrasound was implemented by the therapist. The ultrasound parameters were set as following, frequency: 1 MHz, intensity: 0.5 W/cm2 and the treatment time was 5 minutes
  Interventions: Combination Product: phonophoresis with different material

INTERVENTIONS:
Combination Product: phonophoresis with different material — phonophoresis with Silicone gel for group A, , Group B: 15 patients (8 males and 7 females) received phonophoresis with Contractubex gel and Group C: 15 patients (9 males and 6 females) received Corticosteroid phonophoresis.

SUMMARY:
Hypertrophic scars and keloids are physically and mentally disturbed, and in addition, can cause pain and itching. Various treatment is utilized to diminish or counteract scarring. The purpose of this study was conducted to compare the effect of Silicone gel, Contractubex gel and Corticosteroid Phonophoresis for Post-burn Hypertrophic Scars. Forty-five patients with hypertrophic scars after 2 to 4 months post thermal burn, their age groups ranged from 20-45 years. Patients were randomly assigned to three groups; Group A: 15 patients (8 males and 7 females) received phonophoresis with Silicone gel, Group B: 15 patients (8 males and 7 females) received phonophoresis with Contractubex gel and Group C: 15 patients (9 males and 6 females) received Corticosteroid phonophoresis. All treatment interventions were applied at a frequency of 3sessions /week for 24 weeks. Outcome measures were performed through modified Vancouver scar scale. The assessment was done pretreatment, after 12 weeks and after 24 weeks of the treatment.

DETAILED DESCRIPTION:
Participants A convenient sample of forty-five patients, 25 male and 20 female, were recruited from the Outpatient Clinic Kasr El-Ani hospital to be treated in the Outpatient Clinic, Faculty of Physical Therapy, Cairo University. They were enrolled and assessed for their eligibility to participate in the study. To be included in the study, patients had hypertrophic scars after 2 to 4 months post thermal burn (direct flame or scald) all patients injury was deep second-degree burn and their age ranged from 20-45 years, they had been free from any other illness that may affect or impact the results as; skin disease, diabetes, mental disorders, peripheral vascular diseases, acute viral diseases, open wound, electrical and chemical burns were excluded.

Randomization Informed consent was obtained from each participant after explaining the nature, purpose, and benefits of the study, informing them of their right to refuse or withdraw at any time, and about the confidentiality of any obtained information. Anonymity was assured through coding of all data. Participants with hypertrophic scar post burn were randomly assigned into three groups (group A, group B and group C) by a blinded and an independent research assistant who opened sealed envelopes that contained a computer-generated randomization card. No subjects dropped out of the study after randomization.

Interventions Participants were randomly assigned into group A (GA) received Silicone gel phonophoresis: Silicone gel (strataderm) was applied to the scar then the ultrasound was implemented by the therapist. The ultrasound parameters were set as following, frequency: 1 MHz, intensity: 0.5 W/cm2 and the treatment time was 5 minutes. The Ultrasound Device is Sonopulse 590: Nonius, sonopuls 590, S.NO.03-202 type 14663.900 was a therapeutic ultrasound device manufactured by Enraf Holland.

Group B (GB) received Contractubex phonophoresis: Contractubex (Merz Pharma, Frankfurt, Germany was applied to the scar then the ultrasound was implemented by the therapist. The ultrasound parameters were set as following, frequency: 1 MHz, intensity: 0.5 W/cm2 and the treatment time was 5 minutes.

Group C (GC) received Corticosteroid phonophoresis: A thin film of coupling medium (gel) was put on the hypertrophic scar and sufficient quantity of Triamcinolone was put by a syringe over the whole scar then the ultrasound was implemented by the therapist. The ultrasound parameters were set as following, frequency: 1 MHz, intensity: 0.5 W/cm2 and the treatment time was 5 minutes. All groups received 72 sessions of treatment, three times per week for 24 weeks.

Outcome measures Scar assessment was done using the modified Vancouver scar scale (Danielsen et al., 2013). The modified scale is a numerical assessment of four skin characteristics, where 0 represents the person's normal skin. The characteristics include height (range 0-3), pliability (range 0-5), vascularity (range 0-3), and pigmentation (range 0-3). The assessment was done before treatment, after three months (12 weeks) (post 1) and after six months (24 weeks) of the treatment (post 2). The final outcome was measured after six months of follow-up, in terms of complete and incomplete recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients had hypertrophic scars after 2 to 4 months post thermal burn (direct flame or scald) all patients injury was deep second-degree burn and their age ranged from 20-45 years

Exclusion Criteria:

* skin disease, diabetes, mental disorders, peripheral vascular diseases, acute viral diseases, open wound, electrical and chemical burns were excluded

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
change of modified Vancouver scar scale | pretreatment, after 12 weeks and after 24 weeks of the treatment
  Scar assessment was done using the modified Vancouver scar scale (Danielsen et al., 2013). The modified scale is a numerical assessment of four skin characteristics, where 0 represents the person's normal skin. The characteristics include height (range 0-3), pliability (range 0-5), vascularity (range 0-3), and pigmentation (range 0-3). The assessment was done before treatment, after three months (12 weeks) (post 1) and after six months (24 weeks) of the treatment (post 2). The final outcome was measured after six months of follow-up, in terms of complete and incomplete recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Hamada A Hamada, Principal Investigator — Cairo University
Locations (1):
- Hamada Ahmed Hamada, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sinha S, Gabriel VA, Arora RK, Shin W, Scott J, Bharadia SK, Verly M, Rahmani WM, Nickerson DA, Fraulin FO, Chatterjee P, Ahuja RB, Biernaskie JA. Interventions for postburn pruritus. Cochrane Database Syst Rev. 2024 Jun 5;6(6):CD013468. doi: 10.1002/14651858.CD013468.pub2. PMID 38837237